CLINICAL TRIAL: NCT06861491
Title: Student Pharmacist Intervention on Type 2 Diabetes Management in Older Adult Populations
Brief Title: Student Pharmacist Non-Pharmacological Intervention on Type 2 Diabetes Management in Older Asian Adult Populations
Acronym: SPY-DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-42131
Record Dates: First submitted 2025-02-17; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: student pharmacist; non-pharmacological; diabetes; management; SPY-DM; glucose control; Asian; Older adult
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-pharmacological intervention and education by student pharmacists (Experimental): Student pharmacists will provide non-pharmacological recommendations to participants about lifestyle modifications, including exercise and diet, as well as provide information about current medications the participant is taking.
  Interventions: Behavioral: Non-pharmacological
- Control (No Intervention): Student pharmacists will collect data on participants, but will not provide recommendations on non-pharmacological management. However, they will provide online resources on diabetes management if prompted.

INTERVENTIONS:
Behavioral: Non-pharmacological — This intervention will be provided by student pharmacists. It will focus on lifestyle modifications, adherence, and education of disease state.
  Other Names: Lifestyle; Diet; Exercise; Adherence
  Arms: Non-pharmacological intervention and education by student pharmacists

SUMMARY:
This study is being done to assess the impact of student pharmacist involvement on blood glucose control through non-pharmacological interventions in people of Asian and Asian descent over the age of 50 with type 2 diabetes. This study team is trying to advance the field of pharmacy and expand the roles of student pharmacists.

DETAILED DESCRIPTION:
This study aims to assess the clinical impact of student pharmacist-led interventions on glycemic control in adult populations. This study will specifically target adults aged 50 years and older of Asian or Asian-descent with diagnosed type 2 diabetes, residing in San Francisco. The goal of the study is to demonstrate the utility of pharmacy students in a community setting on chronic disease management through patient-specific education and interventions. The aims of this study are to compare glycemic control in patients with type 2 diabetes who receive continuous assessment and non-pharmacological counseling from student pharmacists versus those who do not. Specifically, this study will evaluate:

1. The impact of student pharmacist assessments and personalized recommendations on diet, exercise, and adherence to treatment regimens, and their lasting effects on blood glucose control.
2. If participants perceived any value and effect of student pharmacist involvement in managing chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 50 years old
* Asian or Asian-descent
* Diagnosed with T2DM
* A1C >7.0% (uncontrolled)
* Take blood glucose measurements as prescribed by their physician, or consistently (defined as missing no more than 1 reading from their regular routine).

Exclusion Criteria:

* Age < 50 years old
* Not diagnosed with type 2 diabetes, or have diagnoses such as type 1 diabetes, gestational diabetes, or medication induced diabetes
* Patients that are on medications that affect glycemic control
* Corticosteroids
* First-generation antipsychotics (e.g. chlorpromazine, perphenazine, phenothiazines)
* Immunosuppressants (e.g. tacrolimus, cyclosporine)
* Experiencing acute disease states
* Recent surgery/hospitalized within the last 3 months
* Active infections
* Non-adherence to blood glucose monitoring (defined as missing > 1 reading from their regular routine or not taking readings as prescribed by their doctor)
* Patients with late stage T2DM requiring insulin therapy
* Diagnosed with cancer, end-stage renal disease, end-stage liver disease
* Received any organ transplant

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Blood glucose control | Up to 12 months
  This will assess the average blood glucose change over the course of the study.
A1C | Up to 12 months
  To assess effect of student pharmacist non-pharmacological intervention on A1C levels

SECONDARY OUTCOMES:
Utilization of Questionnaires to assess Comprehension of Diabetes Management | Up to 12 months
  Student pharmacists will be assessed on their change in understanding of type 2 diabetes management through an assessment that will be scored. Study participants will also be assessed on their comfort and understanding of type 2 diabetes as a disease state, as well as basic management through a form that will be scored.
  Once the questionnaire is finalized, participants will be asked to complete the form with higher scores indicating better level of understanding.
Utilization of Questionnaires to assess Participant Perceptions of Student Pharmacist Involvement on Chronic Disease Management | Up to 12 months
  Study participants will be asked to complete a questionnaire to reflect on their experiences with student pharmacists. Overall perception of their experience will be collected utilizing a combination of short-answer and multiple-choice questions. Multiple-choice questions will be analyzed using Likert Scale with higher values representing favorable outcomes. Short-answer questions will be coded to identify overall themes of the study to address areas for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Zhou, PharmD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No